CLINICAL TRIAL: NCT03034915
Title: A 24-week Treatment, Multi-center, Randomized, Double-blind, Double-dummy, Parallel Group Study to Compare Umeclidinium/Vilanterol, Umeclidinium, and Salmeterol in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A 24-week Study to Compare Umeclidinium/Vilanterol (UMEC/VI), UMEC and Salmeterol in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201749; 2016-002513-22 (EudraCT Number)
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Vilanterol; COPD; HRQoL; Salmeterol; Umeclidinium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- UMEC/VI 62.5/25 mcg via ELLIPTA + placebo via DISKUS (Experimental): Subjects will be instructed to self-administer one dose of UMEC/VI 62.5/25 mcg inhalation powder each morning via ELLIPTA DPI and placebo twice daily (morning and evening) via DISKUS DPI.
  Interventions: Drug: UMEC/VI 62.5/25 mcg via ELLIPTA; Drug: Placebo via DISKUS
- UMEC 62.5 mcg via ELLIPTA + placebo via DISKUS (Experimental): Subjects will be instructed to self-administer one dose of UMEC 62.5 mcg inhalation powder each morning via ELLIPTA DPI and placebo twice daily (morning and evening) via DISKUS DPI.
  Interventions: Drug: UMEC 62.5 mcg via ELLIPTA; Drug: Placebo via DISKUS
- Salmeterol 50 mcg via DISKUS + placebo via ELLIPTA (Experimental): Subjects will be instructed to self-administer one dose of salmeterol 50 mcg twice daily (morning and evening) via DISKUS DPI and placebo once daily morning via ELLIPTA DPI.
  Interventions: Drug: Salmeterol 50 mcg via DISKUS; Drug: Placebo via ELLIPTA

INTERVENTIONS:
Drug: UMEC/VI 62.5/25 mcg via ELLIPTA — ELLIPTA DPI inhaler will contain two individual blister strips with 30 blisters per strip; the first strip contains umeclidinium bromide (62.5 mcg per blister) blended with lactose monohydrate and magnesium stearate and second strip contains vilanterol trifenatae (25 mcg per blister) blended with lactose monohydrate and magnesium stearate.
  Arms: UMEC/VI 62.5/25 mcg via ELLIPTA + placebo via DISKUS
Drug: UMEC 62.5 mcg via ELLIPTA — The ELLIPTA inhaler will contain one blister strip, which will have 30 blisters of umeclidinium bromide (62.5 mcg).
  Arms: UMEC 62.5 mcg via ELLIPTA + placebo via DISKUS
Drug: Salmeterol 50 mcg via DISKUS — The DISKUS inhaler will contain one blister strip, which will have 60 blisters of salmeterol xinafoate (50 mcg). The DISKUS will provide a total of 60 doses (60 blisters) and will deliver, when actuated, the contents of a single blister strip.
  Arms: Salmeterol 50 mcg via DISKUS + placebo via ELLIPTA
Drug: Placebo via ELLIPTA — Lactose dry powder will be administered using ELLIPTA for both treatment periods. ELLIPTA DPI inhaler will contain two individual blister strips with 30 blisters per strip; containing lactose dry powder.
  Arms: Salmeterol 50 mcg via DISKUS + placebo via ELLIPTA
Drug: Placebo via DISKUS — Lactose dry powder will be administered using DISKUS for both treatment periods. The DISKUS inhaler will contain one blister strip, which will have 60 blisters of lactose dry powder. The DISKUS will provide a total of 60 doses (60 blisters) and will deliver, when actuated, the contents of a single blister strip.
  Arms: UMEC 62.5 mcg via ELLIPTA + placebo via DISKUS; UMEC/VI 62.5/25 mcg via ELLIPTA + placebo via DISKUS

SUMMARY:
COPD is characterized by an airflow limitation, which is not fully reversible, usually progressive and accompanied by chronic cough, sputum production and dyspnea, which can be a major cause of disability and anxiety associated with the disease. In addition, COPD is associated with poor health-related quality of life (HRQoL). Pharmacologic therapy is used to improve lung function, reduce symptoms, reduce the frequency and severity of exacerbations, and also to improve health status and exercise tolerance.

This is a multi-center, randomized, double blind, double dummy, 3-arm parallel group study to compare umeclidinium/vilanterol (62.5/25 microgram [mcg], once daily), umeclidinium (62.5 mcg, once daily), and salmeterol (50 mg, twice daily) in male and female subjects with COPD. The primary purpose of this study is to demonstrate improvements in lung function for subjects treated with UMEC/VI compared with UMEC for 24 weeks.

Approximately 2424 subjects will be randomized across 3 parallel arms in 1:1:1 ratio. Subjects will be stratified based on long-acting bronchodilator usage during the run-in period (none, one or 2 long-acting bronchodilators per day). Subjects will receive either UMEC/VI inhalation powder (62.5/25 microgram [mcg] once daily) administered via the ELLIPTA® dry powder inhaler (DPI) and placebo twice daily via DISKUS® DPI; or UMEC (62.5 mcg once daily) administered via the ELLIPTA DPI and placebo twice daily via DISKUS DPI or salmeterol (50 mcg twice daily [BID]) administered via the DISKUS DPI and placebo once daily via ELLIPTA DPI. The duration of the study will be 29 to 31 weeks including a pre-screening period of 2 weeks, run-in period of 4 weeks, treatment period of 24 weeks and follow-up period of 1 week.

ELLIPTA and DISKUS are trademarks of GSK group of companies.

ELIGIBILITY:
Inclusion Criteria

* 40 years or older at date of signing informed consent at Screening Visit 1
* Outpatient with a diagnosis of COPD
* Persistent airflow limitations as indicated by a pre and post-albuterol/salbutamol FEV1/FVC ratio of <0.70 and a post-albuterol/salbutamol FEV1 of >=30% to <=80% predicted normal values at Screening Visit 1.
* A CAT score of >=10 at Screening Visit 1
* Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years (number of pack years = [number of cigarettes per day / 20] multiplied by number of years smoked [e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years both equal 10 pack-years]). Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Pipe and/or cigar use cannot be used to calculate pack-year history.
* Male and female subjects are eligible to participate in the study. A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin test), not lactating, and at least one of the following conditions applies: non-reproductive potential defined as pre-menopausal females with documented tubal ligation or documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or hysterectomy or documented bilateral oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases, a blood sample with simultaneous follicle stimulating hormone and estradiol levels consistent with menopause must be tested. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

A female subject with reproductive potential is eligible to participate if she is not pregnant and agrees to follow one of the highly effective methods for avoiding pregnancy in females of reproductive potential from 30 days prior to the first dose of study medication and until (at least five terminal half-lives or until any continuing pharmacologic effect has ended, whichever is longer) after the last dose of study medication and completion of the follow-up visit. The investigator is responsible for ensuring that subjects understand how to properly use methods of contraception.

* Capable of giving signed informed consent prior to study participation.

Exclusion criteria

* A current diagnosis of asthma (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD, which is the primary cause of their respiratory symptoms).
* Subjects with known alpha-antitrypsin deficiency as the underlying cause of COPD
* Subjects with active tuberculosis are excluded. Subjects with other respiratory disorders (e.g., clinically significant: bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases) are excluded if these conditions are the primary cause of their respiratory symptoms.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease as per investigator assessment); stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice, or cirrhosis; chronic stable hepatitis B and C (e.g., presence of hepatitis B surface antigen or positive hepatitis C antibody test result or within 3 months prior to first dose of study treatment) are acceptable if subject otherwise meets entry criteria.
* Subjects with unstable or life threatening cardiac disease. The investigational product should be used with caution in subjects with severe cardiovascular disease. In the opinion of the investigator, use will only be considered if the benefit is likely to outweigh the risk in conditions such as myocardial infarction or unstable angina in the last 6 months, or unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months, or New York Heart Association Class IV heart failure.
* The investigator will determine the clinical significance of each abnormal electrocardiogram (ECG) finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. Subjects with the following abnormalities are excluded from participation in the study: atrial fibrillation with rapid ventricular rate >120 beats per minute (bpm), sustained or non-sustained ventricular tachycardia, second degree heart block Mobitz type II or third degree heart block (unless pacemaker or defibrillator had been inserted).
* Subjects with medical conditions such as narrow-angle glaucoma, urinary retention, prostatic hypertrophy, or bladder neck obstruction will be excluded unless, in the opinion of the study physician, the benefit outweighs the risk.
* Any subject who is considered unlikely to survive the duration of the study period or has any rapidly progressing disease or immediate life-threatening illness (e.g., cancer). In addition, any subject who has any other condition (e.g., neurological condition) that is likely to affect respiratory function will not be included in the study.
* Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1. Pneumonia and/or moderate or severe COPD exacerbation that has not resolved at least 14 days prior to Screening Visit 1and at least 30 days following the last dose of oral/systemic corticosteroids (if applicable).
* Subjects who had received inhaled corticosteroids (ICS) or ICS/ long-acting beta-agonist for the treatment of COPD in the 6 weeks prior to Screening Visit1.
* Subjects who had >1 moderate exacerbation in the 12 months prior to Screening Visit 1, or one severe exacerbation requiring hospitalization in the 12 months prior to Screening Visit 1.
* Other respiratory tract infections that have not resolved at least 7 days prior to Screening Visit 1.
* Subjects with lung volume reduction surgery (including procedures such as endobronchial valves) within the 12 months prior to Screening Visit 1.
* Use of long-term oxygen therapy described as resting oxygen therapy >3 Liter (L)/minute (min) at screening required to maintain adequate oxygenation (e.g., oxygen saturation in arterial blood [SaO2] >90%; oxygen use <=3 L/min flow is not exclusionary, and subjects may adjust oxygen levels up or down as needed during the study.)
* Use of ICS within 6 weeks prior to Screening Visit 1; use of depot corticosteroids within 12 weeks prior to Screening Visit 1; use of systemic, oral or parenteral corticosteroids within 6 weeks prior to Screening Visit 1 (Localized corticosteroid injections [e.g., intra-articular and epidural] are permitted); use of antibiotics (for lower respiratory tract infection) within 6 weeks prior to Screening Visit 1; use of phosphodiesterase 4 (PDE4) inhibitor (e.g., roflumilast) within 14 days prior to Screening Visit 1; use of long-acting beta-agonist/ ICS combination products within 6 weeks prior to Screening Visit 1; use of theophyllines within 48 hours prior to Screening Visit 1; use of oral long-acting beta2-agonists within 48 hours and short-acting beta2-agonists within 12 hours prior to Screening Visit 1; use of inhaled short-acting beta2-agonists within 4 hours prior to Screening Visit 1 (use of study provided albuterol/salbutamol is permitted during the study, except in the 4-hour period prior to spirometry testing); use of inhaled short-acting anticholinergics within 4 hours prior to Screening Visit 1; use of inhaled short-acting anticholinergic/short-acting beta2-agonist combination products within 4 hours prior to Screening Visit 1; use of any other investigational medication within 30 days or within 5 drug half-lives (whichever is longer) prior to Screening Visit 1.
* Subject unable to withhold albuterol/salbutamol for the 4-hour period required prior to spirometry testing at each study visit.
* Regular use (prescribed for daily/ regular use, not for as-needed use) of short-acting bronchodilators (e.g., albuterol/salbutamol).
* A known or suspected history of alcohol or drug abuse within 2 years prior to Screening Visit 1 that in the opinion of the investigator would prevent the subject from completing the study procedures.
* Any history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, sympathomimetic, lactose/milk protein or magnesium stearate.
* Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Screening Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Subject is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete questionnaires on the electronic diary.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2696 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (175):
- United States (37):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Lincoln, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, O'Fallon, Illinois
  - GSK Investigational Site, Natchitoches, Louisiana
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, Fridley, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Woodbury, Minnesota
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Monroe, North Carolina
  - GSK Investigational Site, Mooresville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Lancaster, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Sherman, Texas
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Morgantown, West Virginia
- Argentina (20):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Florida, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Lobos, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Paraná, Buenos Aires
  - GSK Investigational Site, Quilmes, Buenos Aires
  - GSK Investigational Site, Vicente López, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Concepción del Uruguay, Entre Ríos Province
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Ciudad Autonoma de Buenis Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Monte Grande
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, Santa Fe
  - GSK Investigational Site, Santa Rosa
- Australia (5):
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Darlinghurst, Sydney, New South Wales
  - GSK Investigational Site, Kanwal, New South Wales
  - GSK Investigational Site, Port Macquarie, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
- Canada (12):
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
- France (4):
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Perpignan
  - GSK Investigational Site, Pessac
- Germany (44):
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Wiesloch, Baden-Wurttemberg
  - GSK Investigational Site, Bamberg, Bavaria
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Peine, Lower Saxony
  - GSK Investigational Site, Wardenburg, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bergisch Gladbach, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Rheine, North Rhine-Westphalia
  - GSK Investigational Site, Warendorf, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Annaberg, Saxony
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Mittweida, Saxony
  - GSK Investigational Site, Teuchern, Saxony-Anhalt
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Schleswig, Schleswig-Holstein
  - GSK Investigational Site, Schmölln, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Leipzig
- Italy (14):
  - GSK Investigational Site, Cassano Delle Murge (BA), Apulia
  - GSK Investigational Site, Benevento, Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Salerno, Campania
  - GSK Investigational Site, San Felice A Cancello (CE), Campania
  - GSK Investigational Site, Reggio Emilia, Emilia-Romagna
  - GSK Investigational Site, Riccione (RN), Emilia-Romagna
  - GSK Investigational Site, Pordenone, Friuli Venezia Giulia
  - GSK Investigational Site, Tradate (VA), Lombardy
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, San Sisto (PG), Umbria
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, San Pietro Vernotico
- Mexico (2):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
- Netherlands (9):
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Beek
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Kloosterhaar
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Zutphen
- South Africa (10):
  - GSK Investigational Site, Eloffsdal, Gauteng
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Middelburg, Mpumalanga
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Panorama
  - GSK Investigational Site, Reiger Park
- Spain (7):
  - GSK Investigational Site, Marbella - Málaga, Andalusia
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Centelles (Barcelona)
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Mérida (Badajoz)
  - GSK Investigational Site, Peralada( Girona)
- Sweden (11):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Höllviken
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Luleå
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Skövde
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20277

REFERENCES:
- [Background] Maltais F, Bjermer L, Kerwin EM, Jones PW, Watkins ML, Tombs L, Naya IP, Boucot IH, Lipson DA, Compton C, Vahdati-Bolouri M, Vogelmeier CF. Efficacy of umeclidinium/vilanterol versus umeclidinium and salmeterol monotherapies in symptomatic patients with COPD not receiving inhaled corticosteroids: the EMAX randomised trial. Respir Res. 2019 Oct 30;20(1):238. doi: 10.1186/s12931-019-1193-9. PMID 31666084
- [Derived] Kerwin EM, Jones PW, Bjermer LH, Maltais F, Boucot IH, Naya IP, Lipson DA, Compton C, Tombs L, Vogelmeier CF. How can the findings of the EMAX trial on long-acting bronchodilation in chronic obstructive pulmonary disease be applied in the primary care setting? Chron Respir Dis. 2023 Jan-Dec;20:14799731231202257. doi: 10.1177/14799731231202257. PMID 37800633
- [Derived] Bjermer LH, Boucot IH, Vogelmeier CF, Maltais F, Jones PW, Tombs L, Compton C, Lipson DA, Kerwin EM. Efficacy and Safety of Umeclidinium/Vilanterol in Current and Former Smokers with COPD: A Prespecified Analysis of The EMAX Trial. Adv Ther. 2021 Sep;38(9):4815-4835. doi: 10.1007/s12325-021-01855-y. Epub 2021 Aug 4. PMID 34347255
- [Derived] Maltais F, Naya IP, Vogelmeier CF, Boucot IH, Jones PW, Bjermer L, Tombs L, Compton C, Lipson DA, Kerwin EM. Salbutamol use in relation to maintenance bronchodilator efficacy in COPD: a prospective subgroup analysis of the EMAX trial. Respir Res. 2020 Oct 22;21(1):280. doi: 10.1186/s12931-020-01451-8. PMID 33092591
- [Derived] Kerwin EM, Boucot IH, Vogelmeier CF, Maltais F, Naya IP, Tombs L, Jones PW, Lipson DA, Keeley T, Bjermer L. Early and sustained symptom improvement with umeclidinium/vilanterol versus monotherapy in COPD: a post hoc analysis of the EMAX randomised controlled trial. Ther Adv Respir Dis. 2020 Jan-Dec;14:1753466620926949. doi: 10.1177/1753466620926949. PMID 32462979

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this randomized, double-blind, double dummy, 3-arm parallel group study, eligible participants received Umeclidinium/Vilanterol (UMEC/VI) 62.5/25 microgram (mcg) once daily via the ELLIPTA dry powder inhaler (DPI), or UMEC 62.5 mcg once daily via ELLIPTA DPI, or Salmeterol (SAL) 50 mcg twice daily (BID) via the DISKUS DPI (1:1:1) for 24 weeks.
Pre-assignment Details: A total of 3591 participants who met the eligibility criteria were screened; 2431 participants were randomized and 2425 comprised the Intent to Treat (ITT) population (6 participants randomized in error and did not receive any treatment).The study consisted of a run-in period (4 weeks), treatment period (24 weeks) and follow up period (7+/-3 days).
Groups:
- UMEC/VI 62.5/25 mcg+ Placebo: Participants with COPD received UMEC/VI 62.5/25 mcg once daily via the ELLIPTA DPI along with placebo twice daily via the DISKUS DPI for 24 weeks. In addition albuterol/salbutamol was provided to participants to use on an as-needed basis for relief of COPD symptoms throughout the study. Participants were followed up 7 days after the last dose of study medication.
- UMEC 62.5 mcg + Placebo: Participants with COPD received UMEC 62.5mcg once daily via the ELLIPTA DPI along with placebo twice daily via DISKUS DPI for 24 weeks. In addition albuterol/salbutamol was provided to participants to use on an as-needed basis for relief of COPD symptoms throughout the study. Participants were followed up 7 days after the last dose of study medication.
- Salmeterol 50 mcg+Placebo: Participants with COPD received salmeterol 50 mcg twice daily via the DISKUS DPI along with placebo once daily via ELLIPTA DPI for 24 weeks. In addition albuterol/salbutamol was provided to participants to use on an as-needed basis for relief of COPD symptoms throughout the study. Participants were followed up 7 days after the last dose of study medication.
Period: Overall Study
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
Started | 812 | 804 | 809
Completed | 717 | 650 | 683
Not Completed | 95 | 154 | 126
Not completed — Adverse Event | 29 | 32 | 22
Not completed — Lost to Follow-up | 5 | 13 | 3
Not completed — Withdrawal by Subject | 29 | 46 | 41
Not completed — Protocol Deviation | 2 | 14 | 7
Not completed — Lack of Efficacy | 8 | 16 | 18
Not completed — Site closed | 2 | 2 | 4
Not completed — Protocol-defined withdrawal criteria met | 19 | 26 | 29
Not completed — Physician Decision | 1 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo | Total
Number analyzed (Participants) | 812 | 804 | 809 | 2425
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (8.37) | 64.9 (8.48) | 64.4 (8.53) | 64.6 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 319 | 327 | 342 | 988
  Male | 493 | 477 | 467 | 1437
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 24 | 23 | 25 | 72
  American Indian or Alaska Native | 13 | 12 | 12 | 37
  Asian - Central/South Asian Heritage | 5 | 0 | 0 | 5
  Asian - Japanese Heritage | 0 | 1 | 0 | 1
  Asian - East Asian Heritage | 0 | 0 | 1 | 1
  White - Arabic/North African Heritage | 3 | 1 | 1 | 5
  White - White/Caucasian/European Heritage | 764 | 763 | 765 | 2292
  American Indian or Alaska Native & White | 1 | 0 | 0 | 1
  Black or African American & White | 2 | 4 | 4 | 10
  Native Hawaiian or other Pacific Islander & White | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) at Week 24
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 at Week 24 is defined as the mean of the FEV1 values obtained 23 and 24 hours after dosing on the previous day. Baseline trough FEV1 is the mean of the values measured at 30 minutes and 5 minutes pre-dose on Day 1. Change from Baseline was calculated as the trough FEV1 value on Week 24 minus the Baseline value. Analysis was performed using a repeated measures model (MMRM) with covariates of Baseline FEV1, geographical region, stratum (number of bronchodilators per day during run-in), visit, treatment, visit by Baseline and visit by treatment interaction. ITT population comprised of all randomized participants (excluding those who were randomized in error) who received at least one dose of study medication.
Time Frame: Baseline (Pre-dose on Day 1) and Week 24
Population: ITT Population. Participants represents those with data available at the time point being presented; however, all participants in the ITT population without missing covariate information and with at least one post Baseline measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
Number analyzed (Participants) | 691 | 621 | 654
Liters | 0.122 (0.0081) | 0.056 (0.0085) | -0.019 (0.0083)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs UMEC 62.5 mcg + Placebo; Test type: Other; p < 0.001, Mixed model repeated measures; Mean Difference (Net) = 0.066, 95% CI 2-sided [0.043 to 0.089], Standard Error of Mean 0.0118 — LS Mean difference comparing UMEC/VI versus UMEC at Week 24
Statistical Analysis 2: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p < 0.001, Mixed model repeated measures; Mean Difference (Net) = 0.141, 95% CI 2-sided [0.118 to 0.164], Standard Error of Mean 0.0117 — LS Mean difference comparing UMEC/VI versus salmeterol at Week 24
Statistical Analysis 3: Comparison: UMEC 62.5 mcg + Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p < 0.001, Mixed model repeated measures; Mean Difference (Net) = 0.075, 95% CI 2-sided [0.051 to 0.098], Standard Error of Mean 0.0119 — LS Mean difference comparing UMEC versus salmeterol at Week 24

2. Secondary Outcome: Self Administered Computerized (SAC) Transient Dyspnea Index (TDI) Focal Score at Week 24
Description: TDI focal score comprises of 3 individual scales (Functional Impairment, Magnitude of Task, Magnitude of Effort). Each of these scales had a possible score ranging from -6 to +6, lower scores indicates impairment. TDI focal score was calculated as the sum of 3 individual scores (range is -18 to +18). Lower score indicates deterioration of dyspnea. If a score is missing for any of the three scales, then the TDI focal score was set to missing. Analysis was performed using mixed model repeated measures (MMRM) with covariates of SAC BDI focal score, geographical region, stratum (no. of bronchodilators per day during run-in), visit, treatment, visit by SAC BDI and visit by treatment interactions.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
Number analyzed (Participants) | 704 | 636 | 673
Scores on a scale | 1.68 (0.109) | 1.30 (0.114) | 1.22 (0.111)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs UMEC 62.5 mcg + Placebo; Test type: Other; p = 0.018, Mixed model repeated measures; Mean Difference (Net) = 0.37, 95% CI 2-sided [0.06 to 0.68], Standard Error of Mean 0.157 — LS Mean difference comparing UMEC/VI versus UMEC at Week 24
Statistical Analysis 2: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.004, Mixed model repeated measures; Mean Difference (Net) = 0.45, 95% CI 2-sided [0.15 to 0.76], Standard Error of Mean 0.155 — LS Mean difference comparing UMEC/VI versus salmeterol at Week 24
Statistical Analysis 3: Comparison: UMEC 62.5 mcg + Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.610, Mixed model repeated measures; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.23 to 0.39], Standard Error of Mean 0.159 — LS Mean difference comparing UMEC versus salmeterol at Week 24

3. Secondary Outcome: Percentage of TDI Responders According to SAC TDI Focal Score
Description: TDI focal score comprises of 3 individual scales (Functional Impairment, Magnitude of Task, Magnitude of Effort). Each of these scales had a possible score ranging from -6 to +6, lower scores indicates impairment. TDI focal score was calculated as the sum of 3 individual scores (range is -18 to +18). Lower score indicates deterioration of dyspnea. If a score is missing for any of the three scales, then TDI focal score was set to missing. A participant was considered as a responder if the on-treatment TDI focal score was at least 1 unit at that visit. Non-response was SAC TDI focal score of less than 1 unit or a missing SAC TDI focal score with no subsequent non-missing on-treatment scores. Analysis was performed using a generalized linear mixed model with treatment as an explanatory variable and visit, SAC BDI focal score, stratum (no. of bronchodilators per day during run-in), geographical region, visit by SAC BDI and visit by treatment interactions included as covariates.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
Number analyzed (Participants) | 806 | 799 | 807
Percentage of responders | 50 | 42 | 41
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs UMEC 62.5 mcg + Placebo; Test type: Other; p < 0.001, generalized linear mixed model; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.17 to 1.75] — Odds Ratio (responder vs. a non-responder) comparing UMEC/VI vs UMEC at Week 24
Statistical Analysis 2: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p < 0.001, generalized linear mixed model; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.21 to 1.81] — Odds Ratio (responder vs. a non-responder) comparing UMEC/VI versus salmeterol at Week 24
Statistical Analysis 3: Comparison: UMEC 62.5 mcg + Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.755, generalized linear mixed model; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.84 to 1.27] — Odds Ratio (responder vs. a non-responder) comparing UMEC versus salmeterol at Week 24

4. Secondary Outcome: Mean Change From Baseline in Evaluating Respiratory Symptoms (E-RS) Total Score
Description: The E-RS is intended to capture information related to respiratory symptoms. A daily symptom score for E-RS is derived by summing 11 item-scores. The domains include: respiratory symptoms (RS)-breathlessness (RS-BRL comprised of 5 items, score range [0-17]), RS-cough and sputum (RS-CSP comprised of 3 items, score range [0-11]), and RS-chest symptoms (RS-CSY comprised of 3 items, score range [0-12]). Total score ranged between 0-40 and higher values indicates severe respiratory symptoms. The instrument was completed each night prior to going to bed. Baseline E-RS score is the mean within-participant daily score over 7 days prior to randomization. Change from Baseline is the difference at Week 21-Week 24 value and Baseline value. Analysis was performed using MMRM with covariates of Baseline score, geographical region, stratum (no. of bronchodilators per day during run-in), 4-weekly period, treatment, 4-weekly period by Baseline and 4-weekly period by treatment interactions.
Time Frame: Baseline (Pre-dose on Day 1) and Week 21 to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
Number analyzed (Participants) | 677 | 621 | 653
Scores on a scale | -1.52 (0.148) | -0.99 (0.152) | -0.69 (0.150)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs UMEC 62.5 mcg + Placebo; Test type: Other; p = 0.013, Mixed model repeated measures; Mean Difference (Net) = -0.53, 95% CI 2-sided [-0.95 to -0.11], Standard Error of Mean 0.213 — LS Mean difference comparing UMEC/VI versus UMEC at Week 21 to Week 24
Statistical Analysis 2: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p < 0.001, Mixed model repeated measures; Mean Difference (Net) = -0.83, 95% CI 2-sided [-1.25 to -0.42], Standard Error of Mean 0.211 — LS Mean difference comparing UMEC/VI versus salmeterol at Week 21 to Week 24
Statistical Analysis 3: Comparison: UMEC 62.5 mcg + Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.159, Mixed model repeated measures; Mean Difference (Net) = -0.30, 95% CI 2-sided [-0.72 to 0.12], Standard Error of Mean 0.214 — LS Mean difference comparing UMEC versus salmeterol at Week 21 to Week 24

5. Secondary Outcome: Mean Change From Baseline in E-RS Subscale Score
Description: as for outcome 4
Time Frame: Baseline (Pre-dose on Day 1) and Week 21 to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
Number analyzed (Participants) | 677 | 621 | 653
Scores on a scale
  RS-BRL | -0.67 (0.080) | -0.40 (0.082) | -0.22 (0.081)
  RS-CSP | -0.45 (0.044) | -0.38 (0.045) | -0.32 (0.044)
  RS-CSY | -0.39 (0.049) | -0.22 (0.050) | -0.15 (0.049)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs UMEC 62.5 mcg + Placebo; Test type: Other; p = 0.016, Mixed model repeated measures — E-RS Breathlessness Score; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.50 to -0.05], Standard Error of Mean 0.114 — LS Mean difference comparing UMEC/VI versus UMEC at Week 21 to Week 24
Statistical Analysis 2: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p < 0.001, Mixed model repeated measures — E-RS Breathlessness Score; Mean Difference (Net) = -0.46, 95% CI 2-sided [-0.68 to -0.23], Standard Error of Mean 0.113 — LS Mean difference comparing UMEC/VI versus salmeterol at Week 21 to Week 24
Statistical Analysis 3: Comparison: UMEC 62.5 mcg + Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.115, Mixed model repeated measures — E-RS Breathlessness Score; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.41 to 0.04], Standard Error of Mean 0.115 — LS Mean difference comparing UMEC versus salmeterol at Week 21 to Week 24
Statistical Analysis 4: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs UMEC 62.5 mcg + Placebo; Test type: Other; p = 0.247, Mixed model repeated measures — E-RS Cough and Sputum Score; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.20 to 0.05], Standard Error of Mean 0.063 — LS Mean difference comparing UMEC/VI versus UMEC at Week 21 to Week 24
Statistical Analysis 5: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.042, Mixed model repeated measures — E-RS Cough and Sputum Score; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.25 to 0.00], Standard Error of Mean 0.063 — LS Mean difference comparing UMEC/VI versus salmeterol at Week 21 to Week 24
Statistical Analysis 6: Comparison: UMEC 62.5 mcg + Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.391, Mixed model repeated measures — E-RS Cough and Sputum Score; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.18 to 0.07], Standard Error of Mean 0.063 — LS Mean difference comparing UMEC versus salmeterol at Week 21 to Week 24
Statistical Analysis 7: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs UMEC 62.5 mcg + Placebo; Test type: Other; p = 0.014, Mixed model repeated measures — E-RS Chest Symptoms Score; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.31 to -0.04], Standard Error of Mean 0.070 — LS Mean difference comparing UMEC/VI versus UMEC at Week 21 to Week 24
Statistical Analysis 8: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p < 0.001, Mixed model repeated measures — E-RS Chest Symptoms Score; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.37 to -0.10], Standard Error of Mean 0.069 — LS Mean difference comapring UMEC/VI versus salmeterol at Week 21 to Week 24
Statistical Analysis 9: Comparison: UMEC 62.5 mcg + Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.340, Mixed model repeated measures — E-RS Chest Symptoms Score; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.20 to 0.07], Standard Error of Mean 0.070 — LS Mean difference comparing UMEC versus salmeterol at Week 21 to Week 24

6. Secondary Outcome: Percentage of E-RS Responders According to E-RS Total Score
Description: The E-RS is intended to capture information related to respiratory symptoms. A daily symptom score for E-RS is derived by summing 11 item-scores. The domains include: RS-BRL comprised of 5 items, score range (0-17); RS-CSP comprised of 3 items, score range (0-11); and RS-CSY comprised of 4 items, score range (0-12). Total score ranged between 0-40 and higher values indicates severe respiratory symptoms. The instrument was completed each night prior to going to bed. Response is defined as an E-RS total score of at least 2 or 3.35 below Baseline. Participants with a Baseline but all missing post-Baseline data are also considered a non-responder. Analysis was performed using a generalized linear mixed model with treatment as an explanatory variable and four-weekly period, Baseline score, stratum (no. of bronchodilators per day during run-in), geographical region, four-weekly period by baseline and four-weekly period by treatment interactions included as covariates.
Time Frame: Week 21 to Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
Number analyzed (Participants) | 809 | 800 | 808
Percentage of responders | 36 | 27 | 27
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs UMEC 62.5 mcg + Placebo; Test type: Other; p < 0.001, generalized linear mixed model; Odds Ratio (OR) = 1.52, 95% CI 2-sided [1.22 to 1.89] — Odds Ratio (responder vs. a non-responder) comparing UMEC/VI vs UMEC at Week 21 to Week 24
Statistical Analysis 2: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p < 0.001, generalized linear mixed model; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.23 to 1.90] — Odds Ratio (responder vs. a non-responder) comparing UMEC/VI versus salmeterol at Week 21 to Week 24
Statistical Analysis 3: Comparison: UMEC 62.5 mcg + Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.969, generalized linear mixed model; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.80 to 1.26] — Odds Ratio (responder vs. a non-responder) comparing UMEC versus salmeterol at Week 21 to Week 24

7. Secondary Outcome: Change From Baseline in St George's Respiratory Questionnaire (SGRQ) Total Score
Description: SGRQ is a disease-specific questionnaire designed to measure impact of respiratory disease and its treatment on HRQoL of participants with COPD. It contains 14 questions with a total of 40 items grouped into domains (Symptoms, Activity and Impacts). SGRQ total score was calculated as 100 multiplied by summed weights from all positive items divided by sum of weights for all items in questionnaire. It ranges from 0 to 100, higher score indicates poor HRQoL. Baseline is last non-missing score recorded prior to dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the value at Week 24. Analysis was performed using mixed model repeated measures (MMRM) with covariates of Baseline SGRQ total score, geographical region, stratum (no. of bronchodilators per day during run-in), visit, treatment, visit by Baseline and visit by treatment interactions.
Time Frame: Baseline (Pre-dose on Day 1) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
Number analyzed (Participants) | 704 | 636 | 674
Scores on a scale | -4.98 (0.465) | -5.23 (0.484) | -3.29 (0.475)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs UMEC 62.5 mcg + Placebo; Test type: Other; p = 0.709, mixed model repeated measure; Mean Difference (Net) = 0.25, 95% CI 2-sided [-1.07 to 1.57], Standard Error of Mean 0.672 — LS Mean difference comparing UMEC/VI versus UMEC at Week 24
Statistical Analysis 2: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.011, mixed model repeated measure; Mean Difference (Net) = -1.69, 95% CI 2-sided [-2.99 to -0.39], Standard Error of Mean 0.665 — LS Mean difference comparing UMEC/VI versus salmeterol at Week 24
Statistical Analysis 3: Comparison: UMEC 62.5 mcg + Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.004, mixed model repeated measure; Mean Difference (Net) = -1.94, 95% CI 2-sided [-3.27 to -0.61], Standard Error of Mean 0.678 — LS Mean difference comparing UMEC versus salmeterol at Week 24

8. Secondary Outcome: Percentage of Responders Based on the Saint (St) George Respiratory Questionnaire COPD Specific (SGRQ) Total Score
Description: SGRQ is a disease-specific questionnaire designed to measure impact of respiratory disease and its treatment on HRQoL of participants with COPD. It contains 14 questions with a total of 40 items grouped into domains (Symptoms, Activity and Impacts). SGRQ total score was calculated as 100 multiplied by summed weights from all positive items divided by sum of weights for all items in questionnaire. It ranges from 0 to 100, higher score indicates poor HRQoL. Analysis was performed using a generalized linear mixed model with treatment as an explanatory variable and visit, Baseline SGRQ score, stratum (no. of bronchodilators per day during run-in), geographical region, visit by Baseline and visit by treatment interactions included as covariates. Response was defined as an SGRQ total score of 4 or more units below Baseline.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
Number analyzed (Participants) | 811 | 802 | 809
Percentage of responders | 45 | 41 | 36
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs UMEC 62.5 mcg + Placebo; Test type: Other; p = 0.063, generalized linear mixed model; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.99 to 1.48] — Odds Ratio (responder vs. a non-responder) comparing UMEC/VI versus UMEC at Week 24
Statistical Analysis 2: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p < 0.001, generalized linear mixed model; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.22 to 1.83] — Odds Ratio (responder vs. a non-responder) comparing UMEC/VI versus salmeterol at Week 24
Statistical Analysis 3: Comparison: UMEC 62.5 mcg + Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.045, generalized linear mixed model; Odds Ratio (OR) = 1.23, 95% CI 2-sided [1.00 to 1.51] — Odds Ratio (responder vs. a non-responder) comparing UMEC versus salmeterol at Week 24

9. Secondary Outcome: Change From Baseline in COPD Assessment Test (CAT)
Description: The CAT is a participant-completed instrument designed to provide a simple and reliable measure of health status in COPD for the assessment and long-term follow-up of the individual participant. The CAT consists of eight items, each formatted on a differential scale. Participants rated their experience on a 6-point scale for each question, ranging from 0 (no impact) to 5 (high impact). A total CAT score was calculated by summing the non-missing scores on the eight items ranging from 0 to 40 with higher scores indicating greater disease impact. Baseline is defined as the last non-missing score recorded prior to dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the value at Week 24. Analysis was performed using mixed model repeated measures (MMRM) with covariates of Baseline CAT score, geographical region, stratum (no. of bronchodilators per day during run-in), visit, treatment, visit by Baseline and visit by treatment interactions.
Time Frame: Baseline (Pre-dose on Day 1) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
Number analyzed (Participants) | 703 | 633 | 669
Scores on a scale | -3.5 (0.21) | -3.4 (0.22) | -2.9 (0.21)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs UMEC 62.5 mcg + Placebo; Test type: Other; p = 0.891, mixed model repeated measures; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.6 to 0.6], Standard Error of Mean 0.30 — LS Mean difference comparing UMEC/VI versus UMEC at Week 24
Statistical Analysis 2: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.074, mixed model repeated measures; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.1 to 0.1], Standard Error of Mean 0.30 — LS Mean difference comparing UMEC/VI versus salmeterol at Week 24
Statistical Analysis 3: Comparison: UMEC 62.5 mcg + Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.107, mixed model repeated measures; Odds Ratio (OR) = -0.5, 95% CI 2-sided [-1.1 to 0.1], Standard Error of Mean 0.31 — LS Mean difference comparing UMEC versus salmeterol at Week 24

10. Secondary Outcome: Percentage of Responders According to CAT
Description: The CAT is a participant-completed instrument designed to provide a simple and reliable measure of health status in COPD for the assessment and long-term follow-up of the individual participant. The CAT consists of eight items. Participants rated their experience on a 6-point scale for each question, ranging from 0 (no impact) to 5 (high impact). A total CAT score was calculated by summing the non-missing scores on the eight items ranging from 0 to 40 with higher scores indicate greater disease impact. Response was defined as an CAT score of >=2 below Baseline. Non response was defined as CAT score <2 units below Baseline or a missing CAT score with no subsequent on treatment scores. Analysis performed using a generalized linear mixed model with treatment as an explanatory variable and visit, baseline CAT score, stratum (no. of bronchodilators per day during run-in), geographical region, visit by baseline and visit by treatment interactions included as covariates.
Time Frame: Week 24
Population: ITT Population.
Measure: Number; unit: Percentage of responders
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
Number analyzed (Participants) | 812 | 804 | 809
Percentage of responders | 55 | 48 | 50
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs UMEC 62.5 mcg + Placebo; Test type: Other; p = 0.003, generalized linear mixed model; Odds Ratio (OR) = 1.35, 95% CI 2-sided [1.11 to 1.65] — Odds Ratio (responder vs. a non-responder) comparing UMEC/VI versus UMEC at Week 24
Statistical Analysis 2: Comparison: UMEC/VI 62.5/25 mcg+ Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.037, generalized linear mixed model; Odds Ratio (OR) = 1.23, 95% CI 2-sided [1.01 to 1.50] — Odds Ratio (responder vs. a non-responder) comparing UMEC/VI versus salmeterol at Week 24
Statistical Analysis 3: Comparison: UMEC 62.5 mcg + Placebo vs Salmeterol 50 mcg+Placebo; Test type: Other; p = 0.363, generalized linear mixed model; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.75 to 1.11] — Odds Ratio (responder vs. a non-responder) comparing UMEC versus salmeterol at Week 24

11. Secondary Outcome: Number of Participants With on Treatment Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant , temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events associated with liver injury and impaired liver function based on pre-defined criteria were categorized as SAE.
Time Frame: Up to Week 24
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
Number analyzed (Participants) | 812 | 804 | 809
Participants
  Any AE | 315 | 316 | 314
  Any SAE | 49 | 35 | 38

ADVERSE EVENTS:
Time Frame: On-Treatment serious adverse events (SAEs) and non-serious AEs (nSAEs) were collected from start of study treatment until Week 24.
Description: On-Treatment SAEs and nSAEs were reported for ITT Population.
Arm/Group | UMEC/VI 62.5/25 mcg+ Placebo | UMEC 62.5 mcg + Placebo | Salmeterol 50 mcg+Placebo
All-Cause Mortality (participants affected / at risk) | 4/812 | 4/804 | 0/809
Serious Adverse Events (participants affected / at risk) | 49/812 | 35/804 | 38/809
Other Adverse Events (participants affected / at risk) | 68/812 | 87/804 | 84/809
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UMEC/VI 62.5/25 mcg+ Placebo (N=812) | UMEC 62.5 mcg + Placebo (N=804) | Salmeterol 50 mcg+Placebo (N=809)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7) | 9 (9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 4 (4) | 5 (5)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Muscle abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (2) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post-thoracotomy pain syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Basilar artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tethered cord syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UMEC/VI 62.5/25 mcg+ Placebo (N=812) | UMEC 62.5 mcg + Placebo (N=804) | Salmeterol 50 mcg+Placebo (N=809)
Nasopharyngitis (Infections and infestations) | 68 (81) | 87 (103) | 84 (94)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT03034915/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT03034915/SAP_001.pdf